CLINICAL TRIAL: NCT04279626
Title: The Surgical Outcome of Two-port Laparoscopic Myomectomy Using Conventional Laparoscopic Instruments and Glove-port Technique
Brief Title: Surgical Outcome of Two-port Laparoscopic Myomectomy
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202001027RINA
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Uterine Myoma
Keywords: Laparoscopy; Two-port
MeSH Terms: conditions — Myofibroma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LETS-M: Women who were older than 20 years old and had not reached menopause, with symptomatic uterine myomas, such as hypermenorrhea, infertility, a mass effect-related urinary frequency, and constipation, received LETS-M.
  Interventions: Procedure: LETS-M

INTERVENTIONS:
Procedure: LETS-M — A 1.5-centimeter skin incision was made over the umbilicus, and the abdominal wall was opened layer by layer with an open method. A wound retractor (Alexis, 2-4 centimeter; Applied Medical Resources Corp., Rancho Santa Margarita, CA) was placed, and the glove port was set up, with a 10-millimeter trocar in the thumb over patient's right side, and a 5-millimeter trocar in the little finger over the left side. The pneumoperitoneum was established. A 10-millimeter rigid laparoscope was inserted via the 10-millimeter trocar and controlled by the assistant. The ancillary 5-millimeter port was made over the left lower abdomen under laparoscope inspection. The surgeon performed the surgery via the two 5-millimeter trocars.

SUMMARY:
Study Objective: To evaluate the surgical outcome of laparoendoscopic two-sites myomectomy (LETS-M) and compare the difference between an experienced surgeon and three trainees.

Design: A retrospective study. Setting: A university hospital and a tertiary care center. Patients: 204 women underwent LETS-M

DETAILED DESCRIPTION:
Laparoscopic myomectomy (LM) is an alternative and advanced technique that can take the place of traditional open surgery and achieve the goal of minimally invasive operation for women who wish to preserve the uterus. However, LM is considered a time-consuming procedure, requiring more suturing and knot-tying, and is better performed for woman with an appropriate uterine size by experienced surgeons.

Laparoendoscopic two-sites myomectomy (LETS-M) is a novel setting for LM on a two-port basis, using the umbilical glove port, three trocars, and conventional laparoscopic equipment.

Between January 2015 and September 2019, the medical records of women with uterine myoma managed by LETS-M were retrospectively reviewed.

The review of the chart records consisted of a detailed history, such as age, body mass index (BMI), gravidity, parity, marital status, sexual experience, previous abdominal surgery, and hospital stay after the surgery. All women received preoperative ultrasound for their uterine myoma assessment, including the location, type, size, number, and accompanying pathology, such as an ovarian tumor. The myoma locations were identified during the operation and classified into fundal wall myoma, anterior wall myoma, posterior wall myoma, and cervical myoma. The myoma type classification was based on the International Federation of Gynecology and Obstetrics (FIGO) leiomyoma subclassification system. We measured the weight of the specimen after finishing the surgery. The operation time was defined as the period from the incision to the closure of the skin. Any intraoperative blood loss less than 50mL or minimal blood loss on operation note was recorded as 50 milliliters in this study. Excessive blood loss was defined as more or equal to 500 milliliters in the operation. The postoperative pain scale was evaluated by a visual analog scale (VAS) on the first and second postoperative days.

ELIGIBILITY:
Inclusion Criteria:

* Women older than 20 years old and had not reached menopause
* Symptomatic uterine myomas, such as hypermenorrhea, infertility, a mass effect-related urinary frequency, and constipation.

Exclusion Criteria:

* Dominant symptoms with active pelvic or urinary tract infection
* A history of pelvic radiotherapy
* A preexisting or suspicious malignant pelvic tumor
* Pathologies other than uterine myoma noted during the operation

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women who were older than 20 years old and had not reached menopause, with symptomatic uterine myomas, such as hypermenorrhea, infertility, a mass effect-related urinary frequency and constipation, received LETS-M for their uterine myoma.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Operation time | 1 day (the operation day)
  The operation time was defined as the period from the incision to the closure of the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chun Chang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and analyzed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Result] Lee D, Lee JR, Suh CS, Kim SH. A systematic review and meta-analysis comparing single port laparoscopic myomectomy with conventional laparoscopic myomectomy. Eur J Obstet Gynecol Reprod Biol. 2019 Aug;239:52-59. doi: 10.1016/j.ejogrb.2019.06.001. Epub 2019 Jun 3. PMID 31181399
- [Result] Stewart EA. Uterine fibroids. Lancet. 2001 Jan 27;357(9252):293-8. doi: 10.1016/S0140-6736(00)03622-9. PMID 11214143
- [Result] Chang WC, Huang SC, Sheu BC. Advances in gynecological laparoscopic surgery. J Formos Med Assoc. 2010 Apr;109(4):245-7. doi: 10.1016/s0929-6646(10)60049-6. No abstract available. PMID 20440899
- [Result] Kim YW, Park BJ, Ro DY, Kim TE. Single-port laparoscopic myomectomy using a new single-port transumbilical morcellation system: initial clinical study. J Minim Invasive Gynecol. 2010 Sep-Oct;17(5):587-92. doi: 10.1016/j.jmig.2010.04.009. Epub 2010 Jun 23. PMID 20576473
- [Result] Munro MG, Critchley HO, Broder MS, Fraser IS; FIGO Working Group on Menstrual Disorders. FIGO classification system (PALM-COEIN) for causes of abnormal uterine bleeding in nongravid women of reproductive age. Int J Gynaecol Obstet. 2011 Apr;113(1):3-13. doi: 10.1016/j.ijgo.2010.11.011. Epub 2011 Feb 22. PMID 21345435
- [Result] Huang PS, Sheu BC, Huang SC, Chang WC. Intraligamental Myomectomy Strategy Using Laparoscopy. J Minim Invasive Gynecol. 2016 Sep-Oct;23(6):954-61. doi: 10.1016/j.jmig.2016.06.007. Epub 2016 Jun 18. PMID 27327965